CLINICAL TRIAL: NCT03843112
Title: Modulating the Vaginal Microbiome After Implantation Failure A Randomized Placebo Controlled Study of Vaginal Lactobacilli Supplements
Brief Title: Modulating the Vaginal Microbiome After Implantation Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: ARTPred (Unknown); Bifodan A/S (Unknown)
Responsible Party: Principal Investigator, Nicholas Macklon, Professor, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REG-076-2018
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Implantation Failure; Infertility, Female; Vaginal Flora Imbalance
Keywords: Infertility, female; Vaginal microbiome
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: Randomised placebo controlled, double blinded study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigator, care providers and outcome assessors are all blinded until the end of inclusion af the last subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vivag Plus (Active Comparator): Vivag Plus vaginal supplements one capsule every night for ten days start cycle day 6-7.
  Interventions: Drug: Vivag Plus
- Placebo (Placebo Comparator): Placebo vaginal supplements one capsule every night for ten days start cycle day 6-7.
  Interventions: Drug: Placebo - Cap

INTERVENTIONS:
Drug: Vivag Plus — Contains two lactobacilli strains; l. gasseri and l. rhamnosus
  Arms: Vivag Plus
Drug: Placebo - Cap — Vaginal supplements
  Other Names: Placebo vaginal capsule
  Arms: Placebo

SUMMARY:
Vaginal microbiome has in studies shown a link with the outcome of fertility treatment. The investigators wish to determine if it is possible to change an unfavorable vaginal microbiome using lactobacilli loaded vaginal supplements.

ELIGIBILITY:
Inclusion Criteria:

* unfavorable vaginal microbiome using ARTPreds test
* non-smoker

Exclusion Criteria:

* use of oral antibiotics oral probiotics between diagnosis and inclusion in the study
* pregnancy at inclusion
* allergy towards study drugs

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-02-27 (Actual)

PRIMARY OUTCOMES:
Change in vaginal microbiome after intervention | 2 months
  The investigators wish to determine if the vaginal microbiome will stay changed one month after intervention. The change in vaginal microbiome will be measured with ARTPreds diagnostic test, after intervention and again one month later. The test divides the vaginal microbiome into three categories, low, medium and high. A change in vaginal microbiome is defined by a shift from low to medium or high, or a shift from medium to high.

CONTACTS AND LOCATIONS:
Locations (1):
- Fertilitetsklinikken, Region Sjælland, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jepsen IE, Saxtorph MH, Englund ALM, Petersen KB, Wissing MLM, Hviid TVF, Macklon N. Probiotic treatment with specific lactobacilli does not improve an unfavorable vaginal microbiota prior to fertility treatment-A randomized, double-blinded, placebo-controlled trial. Front Endocrinol (Lausanne). 2022 Dec 1;13:1057022. doi: 10.3389/fendo.2022.1057022. eCollection 2022. PMID 36531460

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT03843112/Prot_SAP_000.pdf